CLINICAL TRIAL: NCT05405010
Title: Individually Timed Stair Climbing and Descending to Lower Postprandial Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Jeff Moore, Adjunct Professor, San Diego State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: UniquePeakSCD
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Postprandial Hyperglycemia; Postprandial Insulin
MeSH Terms: conditions — Hyperglycemia | interventions — Stair Climbing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Participants remain seated for 1 hour
  Interventions: Other: Seated control
- 1 min (Experimental): Participants remain seated for 1 hour except for 1 minute of stair climbing and descending
  Interventions: Other: Stair climbing and descending for 1 minute
- 3 min (Experimental): Participants remain seated for 1 hour except for 3 minute of stair climbing and descending
  Interventions: Other: Stair climbing and descending for 3 minutes

INTERVENTIONS:
Other: Stair climbing and descending for 1 minute — Stair climbing and descending for 1 minute
  Arms: 1 min
Other: Stair climbing and descending for 3 minutes — Stair climbing and descending for 3 minutes
  Arms: 3 min
Other: Seated control — Seated control
  Arms: Control

SUMMARY:
Effect of individually timed exercise to attenuate postprandial glucose excursions

DETAILED DESCRIPTION:
Participants will perform 1 and 3 minutes stair climbing and descending at a self-selected pace after a mixed meal on separate visits. The timing of these exercise bouts will be determined from an initial control condition where the participant remains seated. Timing of exercise will coincide with the peak glucose from the control condition. Glucose will be measured every 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 years

Exclusion Criteria:

* high-risk from PAR-Q

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Postprandial Glucose | 1 hour
  mg/dL

SECONDARY OUTCOMES:
Postprandial insulin | 1 hour
  iu

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No